CLINICAL TRIAL: NCT02957110
Title: The Relationships Between Laughter Frequency, Pain Perception, and Affect in Fibromyalgia Patients
Brief Title: Laughter Frequency and Fibromyalgia Symptoms
Acronym: LAF
Status: Completed | Type: Observational
Sponsor: Walden University (Other)
Responsible Party: Principal Investigator, Deidre Molchan, Doctoral Student, Walden University
Other Study IDs: 08-05-16-0146047
Record Dates: First submitted 2016-11-02; First posted 2016-11-07 (Estimated); Last update posted 2018-05-07 (Actual); Status verified 2018-05

CONDITIONS: Fibromyalgia
MeSH Terms: conditions — Fibromyalgia

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: Laughter Frequency — Relationships between laughter frequency, momentary mood state, and pain will be observed.

SUMMARY:
The purpose of this study is to investigate whether daily laughter frequency is associated with pain intensity and emotional state ratings in individuals who have fibromyalgia syndrome.

DETAILED DESCRIPTION:
Participants will be asked to provide (or authorize the researcher to obtain) fibromyalgia diagnosis confirmation from a health care provider.

Initially, participants will complete a demographics form and two screening assessments. Then for 14 days, they will be asked to rate their momentary mood and overall pain levels three times per day (shortly after waking up, around 3:00 p.m., and at about an hour before bedtime). At the same time, they will be asked to log each instance of laughter as it occurs, daily, for 14 days. They will carry the log with them throughout each day in order to document each instance of laughter.

ELIGIBILITY:
Inclusion Criteria:

* Individuals who have fibromyalgia syndrome

Exclusion Criteria:

* None.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Individuals who have been diagnosed with fibromyalgia syndrome.
Sampling Method: Non-Probability Sample
Enrollment: 41 (Actual)
Dates: Start 2016-11; Primary Completion 2017-10 (Actual); Study Completion 2017-10 (Actual)

PRIMARY OUTCOMES:
Laughter Frequency | 14 days
  Documenting each instance of laughter throughout each day.
Pain Ratings | Three times per day for 14 days
  Rating overall pain from 0 to 10, three times daily
Emotional State | Three times per day for 14 days
  Rating momentary emotional state three times per day

CONTACTS AND LOCATIONS:
Overall Officials: Ellen Levine, PhD, Study Chair — Walden University
Locations (1):
- Walden University, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No